CLINICAL TRIAL: NCT03718351
Title: Randomized Controlled Trial of Endoscopic Submucosal Dissection Versus Transanal Endoscopic Microsurgery For Early Rectal Neoplasms And Large Rectal Adenomas: Сomparison Of Treatment Efficacy And Safety.
Brief Title: Endoscopic Submucosal Dissection Versus Transanal Endoscopic Microsurgery For Early Rectal Neoplasms And Large Rectal Adenomas: Сomparison Of Treatment Efficacy And Safety.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Principal Investigator, Rybakov Evgeny, MD, Dr. Med. Sc. State Scientific Centre of Coloproctology, Head of Surgical department of oncoproctology, Moscow, Russian Federation, State Scientific Centre of Coloproctology, Russian Federation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104a
Record Dates: First submitted 2018-09-24; First posted 2018-10-24 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Early Rectal Cancer; Large Rectal Adenomas
Keywords: Transanal endoscopic microsurgery; Endoscopic submucosal dissection; Minimally invasive surgery
MeSH Terms: conditions — Rectal Neoplasms | interventions — Transanal Endoscopic Microsurgery; Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transanal endoscopic microsurgery (Active Comparator): a TEM tube will be inserted in the rectum. With specialized instruments the adenoma will be dissected en bloc by a full thickness excision, after which the patient will be admitted to the hospital.
  Interventions: Procedure: transanal endoscopic microsurgery
- endoscopic submucosal dissection (Experimental): an endoscope will be inserted into the rectum and the submucosa underneath the lesion will be injected with saline to lift the adenoma. With an endoscopic knife (Insulated Tip Knife, Olympus or Water Jet, Erbe) the lesion will be resected through the submucosal plane in an eb-bloc fashion, after which the patient will be observed for at least 24h in-hospital.
  Interventions: Procedure: endoscopic submucosal dissection

INTERVENTIONS:
Procedure: transanal endoscopic microsurgery — a TEM tube will be inserted in the rectum. With specialized instruments the adenoma will be dissected en bloc by a full thickness excision, after which the patient will be admitted to the hospital.
  Arms: transanal endoscopic microsurgery
Procedure: endoscopic submucosal dissection — an endoscope will be inserted into the rectum and the submucosa underneath the lesion will be injected with saline to lift the adenoma. With an endoscopic knife (Insulated Tip Knife, Olympus or Water Jet, Erbe) the lesion will be resected through the submucosal plane in an eb-bloc fashion, after which the patient will be observed for at least 24h in-hospital.
  Arms: endoscopic submucosal dissection

SUMMARY:
Transanal endoscopic microsurgery is the main treatment option for rectal tumors such as large adenoma, early cancer because of lower complications and mortality rates and shorter hospital stays rather than conventional surgery. Particularly, However, transanal endoscopic microsurgerymust be performed under either general or spinal anesthesia, and expensive surgical instruments are required. Colorectal endoscopic submucosal dissection is a novel endoscopic procedure that enables en bloc resection of benign colorectal lesions and early colorectal cancer. Endoscopic submucosal dissectioncan be performed under conscious sedation without anesthesia, and there are fewer hospital days than those for transanal endoscopic microsurgery. In the present study, we compared the treatment efficacy and safety between endoscopic submucosal dissectionand transanal endoscopic microsurgery for the treatment of early rectal neoplasms and large rectal adenomas.

ELIGIBILITY:
Inclusion Criteria:

* The lower and upper borders of the adenoma or early rectal cancer are located at ≥2 cm and ≤15 cm from the anal verge, respectively.
* Have signed approved informed consent form for the study
* preoperative stage uT0 and/or uT1, mrT0 and/or mrT1

Exclusion Criteria:

* non-epithelial tumors
* tumors </= 3 cm in size
* recurrent tumors
* suspicion of lymph node metastasis (N + disease)
* preoperative stage uT2 and/or mrT2
* mucous or low-grade adenocarcinoma
* preoperative stage rM1 and/or uM1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-09-24 (Estimated); Study Completion 2021-09-24 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 14 day
En-block resesction rate | 14 day

SECONDARY OUTCOMES:
Incidence of locoregional recurrence | 12 months
Morbidity defined by the Clavien-Dindo classification | 30 day

CONTACTS AND LOCATIONS:
Locations (1):
- State Scientific Centre of Coloproctology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rybakov E, Chernyshov S, Likutov A, Khomiakov E, Yugai O, Alekseev M, Maynovskaia O, Tarasov M, Achkasov S. The results of randomized controlled trial comparing effectiveness of transanal endoscopic microsurgery versus endoscopic submucosal dissection. Surg Endosc. 2026 Jan;40(1):469-474. doi: 10.1007/s00464-025-12319-7. Epub 2025 Oct 24. PMID 41136652